CLINICAL TRIAL: NCT07084987
Title: Effects of Massage, Tub Bathing, and Sponge Bathing on Bilirubin Levels, Skin Barrier, Neonatal Comfort, and Vital Signs: A Randomized Clinical Trial
Brief Title: Massage, Tub Bathing, and Sponge Bathing Effects on Neonatal Bilirubin and Comfort
Acronym: NEO-BATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Rukiye Öztürk, REGİSTERED NURSE, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RUKİYEOZTURK-2025; 2021-42 (Other: Bandırma 17 Eylül University Ethics Committee)
Record Dates: First submitted 2025-07-09; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Hyperbilirubinemia; Newborn Care Phototherapy
Keywords: Neonatal Hyperbilirubinemia; Phototherapy; Neonatal Massage
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of four parallel groups: massage, tub bath, sponge bath, or control.
Masking Description: The study is open-label due to the nature of the interventions, which cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- massage group (Experimental): Newborns receive standardized neonatal massages before phototherapy.
  Interventions: Other: neonatal massage
- Tub Bath Group (Experimental): Newborns receive a warm water tub bath prior to phototherapy.
  Interventions: Other: Tub Bathing
- Sponge Bath Group (Experimental): Newborns receive a sponge (wipe) bath before phototherapy.
  Interventions: Other: sponge bath
- Control Group (No Intervention)

INTERVENTIONS:
Other: neonatal massage — Standardized neonatal massage before phototherapy
  Arms: massage group
Other: Tub Bathing — Tub bath before phototherapy
  Arms: Tub Bath Group
Other: sponge bath — Sponge (wipe) bath before phototherapy
  Arms: Sponge Bath Group

SUMMARY:
This randomized controlled trial evaluates the effects of massage, tub bathing, and sponge bathing on bilirubin levels, skin integrity, neonatal comfort, and physiological parameters in term newborns undergoing phototherapy

DETAILED DESCRIPTION:
Term newborns undergoing phototherapy in the neonatal intensive care unit will be randomized into four groups: massage, sponge bath, tub bath, and control. Pre-intervention assessments include vital signs, skin moisture, bilirubin levels, the Neonatal Comfort Behavior Scale, and the Skin Condition Assessment Scale. Post-intervention assessments are conducted at multiple time points. The study investigates whether massage and bathing interventions can improve comfort, maintain skin integrity, and reduce bilirubin levels more effectively than standard care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion newborns (>37 weeks gestation)

* Receiving phototherapy
* Stable vital signs
* Parental consent

Exclusion Criteria:

* Congenital anomalies
* Severe infections or sepsis
* Parental refusal

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum Bilirubin Levels | Baseline, 6 hours, 24 hours after intervention
  Measured in mg/dL using standard laboratory testing

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye Öztürk, Principal Investigator — Uludag University
Locations (1):
- Bandırma Education and Research Hospital, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect participant privacy and confidentiality.